CLINICAL TRIAL: NCT01769495
Title: A Randomized Trial of the Effect of a Geriatrics Appointment Within 2-3 Days of Discharge From the Emergency Department(ED) in Reducing ED and Hospital Readmissions for Patients 75 Years of Age and Older.
Brief Title: Can a Rapid 2 Day Followup After Discharge From the ED Reduce Readmissions and Death for Patients 75 Years and Older?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: The Duke Endowment (Other); The William R. Kenan, Jr. Charitable Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DE 6366-SP
Record Dates: First submitted 2013-01-14; First posted 2013-01-16 (Estimated); Last update posted 2017-04-17 (Actual); Status verified 2015-04

CONDITIONS: Emergencies
Keywords: Emergency department, Geriatrics, mortality, readmission rates.; Patients 75 years of age and older.
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Standard post ED care
- 2-3 day return appointment (Experimental): Patients will receive further treatment in Geriatric Clinic 2-3 days post ED discharge.
  Interventions: Other: 2-3 day return appointment

INTERVENTIONS:
Other: 2-3 day return appointment — 2-3 appointment in geriatric clinic following ED discharge
  Arms: 2-3 day return appointment

SUMMARY:
Our hypothesis is that a rapid follow up for elderly patients in a Geriatric Clinic discharged from the Emergency Department (ED) will have fewer unplanned return ED visits and fewer unplanned hospital admissions with no attendant increase in mortality.

Patients 75 years of age and older will be randomized following discharge from the ED into two groups. The first will receive standard post ED care. The second will receive an appointment to our Geriatric Clinic within 2-3 days for stabilization, further treatment and contact with the patient's primary physician to communicate the course of the patient's illness and to schedule subsequent follow-up with the patients regular medical provider.

There will be two primary outcomes: The first will be a composite of morality and/or return to the ED at 30 days, and the secondary primary outcome will be mortality. Economic data regarding resource utilization by patients will also be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* All patients 75 years of age and older discharged from the ED

Exclusion Criteria:

* Younger than 75.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 26 (Actual)
Dates: Start 2013-08; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Mortality and readmissions to emergency department | 30 and 180 days

SECONDARY OUTCOMES:
Mortality | 30 and 180 days
  Secondary outcome to measure all cause mortality for patients admitted to the study.

OTHER OUTCOMES:
Medical Resource utilization | 30 days and 180 days

CONTACTS AND LOCATIONS:
Overall Officials: John S Kizer, MD, Principal Investigator — UNC Chapel Hill, NC
Locations (1):
- UNC Hospitals, Chapel Hill, North Carolina, United States